CLINICAL TRIAL: NCT04086758
Title: A Phase 1 Pharmacokinetic Study of Zolbetuximab (IMAB362) in Chinese Subjects With Locally Advanced Unresectable or Metastatic Gastric or Gastro-esophageal Junction (GEJ) Adenocarcinoma
Brief Title: A Pharmacokinetic Study of Zolbetuximab (IMAB362) in Chinese Subjects With Locally Advanced Unresectable or Metastatic Gastric or Gastro-esophageal Junction (GEJ) Adenocarcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma China, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8951-CL-0105
Record Dates: First submitted 2019-09-10; First posted 2019-09-12 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Gastric or Gastro-esophageal Junction (GEJ) Adenocarcinoma
Keywords: Pharmacokinetic; MDV3100; zolbetuximab
MeSH Terms: conditions — Adenocarcinoma | interventions — zolbetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Zolbetuximab (Experimental): Participants will receive a loading dose-1 of zolbetuximab on Day 1 of Cycle 1, consists of 21 days, followed by subsequent lower dose-2 every 3 weeks until they meet the discontinuation criteria.
  Interventions: Drug: zolbetuximab

INTERVENTIONS:
Drug: zolbetuximab — Zolbetuximab will be administered as a 2-hour intravenous infusion
  Other Names: IMAB362

SUMMARY:
A Pharmacokinetic Study of Zolbetuximab (IMAB362) in Chinese Subjects with Locally Advanced Unresectable or Metastatic Gastric or Gastro-esophageal Junction (GEJ) Adenocarcinoma

ELIGIBILITY:
Inclusion Criteria:

* Subject has histologically confirmed diagnosis of gastric or gastro-esophageal junction (GEJ) adenocarcinoma, with radiologically confirmed locally advanced unresectable or metastatic disease, who has no standard of care treatment option or subject is ineligible to receive available standard of care treatment option (any line of treatment).
* Subject agrees not to use another investigational product or medical device while on treatment.
* A female subject is eligible to participate if she is not pregnant (negative serum pregnancy test at screening; female subjects with elevated serum beta human chorionic gonadotropin (βhCG) and a demonstrated non-pregnant status through additional testing are eligible) and at least 1 of the following conditions applies:

  * Not a woman of childbearing potential (WOCBP), OR
  * WOCBP who agrees to follow the contraceptive guidance throughout the treatment period and for at least 6 months after the final study drug administration.
* Female subject must agree not to breastfeed starting at Screening and throughout the study period, and for 6 months after the final study drug administration.
* Female subject must not donate ova starting at screening and throughout the study period, and for 6 months after the final study drug administration.
* A sexually active male subject with female partner(s) who are not of childbearing potential is eligible if:

  * Agree to use a male condom starting at screening and continue throughout study treatment and for 6 months after the final study drug administration.
* A sexually active male subject with female partner(s) who are of childbearing potential must agree to use contraception during the treatment and for at least 6-months after the final study drug administration.
* Male subject must not donate sperm starting at Screening, throughout the study period and for 6 months after the final study drug administration.
* Male subject with a pregnant or breastfeeding partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy or time partner is breastfeeding from the start of screening to 6 months after the final study drug administration.
* Subject has Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Subject has predicted life expectancy ≥ 12 weeks.
* Subject must have an available tumor specimen collected at any time prior to the first dose of study treatment.
* Subject must meet all of the following criteria on the laboratory tests that will be analyzed locally within 14 days prior to the first dose of study drug. In case of multiple laboratory data within this period, the most recent data should be used.

  * Hemoglobin (Hgb) ≥ 9 g/dL (no transfusion within 7 days of start of study treatment)
  * Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L
  * Platelets ≥ 100 × 10^9/L
  * Albumin ≥ 2.5 g/dL
  * Total bilirubin ≤ 1.5 × upper limit of normal (ULN)
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN without liver metastases (≤ 5 x ULN if liver metastases are present)
  * Estimated creatinine clearance ≥ 30 mL/min
  * Prothrombin time/international normalized ratio and partial thromboplastin time ≤ 1.5 × ULN (except for patients receiving anticoagulation therapy)
* Subject's tumor sample has Claudin (CLDN) 18.2 membranous staining in tumor cells with any intensity (≥ 1) as determined by central Immunohistochemistry (IHC) testing.

Exclusion Criteria:

* Subject has prior severe allergic reaction or intolerance to known ingredients of zolbetuximab or other monoclonal antibodies, including humanized or chimeric antibodies like zolbetuximab.
* Subject has received another investigational product or medical device concurrently or within 4 weeks prior first dose of study drug.
* Subject has had radiotherapy within 2 weeks prior to first dose of study treatment. Subject who received palliative radiotherapy to peripheral bone metastases within 2 weeks prior to first dose of study treatment and has recovered from all acute toxicities is allowed.
* Subject has received systemic immunosuppressive therapy, including systemic corticosteroids 2 weeks prior to first dose of study drug. Subjects using a physiologic replacement dose of hydrocortisone or its equivalent (defined as up to 30 mg per day of hydrocortisone or up to 10 mg per day of prednisone) or a single dose of systemic corticosteroid are allowed.
* Subject has gastric outlet obstruction or persistent recurrent vomiting.
* Subject has uncontrolled or significant gastrointestinal hemorrhage.
* Subject has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Subject has a known history of a positive test for human immunodeficiency virus (HIV) infection.
* Subject has a positive test for hepatitis B surface antigen (HBsAg) or hepatitis C virus antibody (anti-HCV). Subjects who are negative for HBsAg, but hepatitis B core antibody (HBcAb) positive, an HB deoxyribonucleic acid (DNA) test will be performed and if positive will be excluded. Subjects with positive serology but negative HCV ribonucleic acid (RNA) test results are eligible.
* Subject has had within 6 months prior to first dose of study treatment any of the following: unstable angina, myocardial infarction, ventricular arrhythmia requiring intervention or hospitalization for heart failure.
* Subject has active infection requiring systemic therapy.
* Subject has clinically significant other disease or co-morbidity, which may adversely affect the safe delivery of treatment within this trial.
* Subject has psychiatric illness or social situations that would preclude study compliance.
* Subject has active autoimmune disease that has required systemic immunosuppressive treatment in the past 2 years.
* Subject has had a major surgical procedure ≤ 28 days prior to the first dose of study drug.

  * Subject has not completely recovered from a major surgical procedure ≤ 14 days prior to the first dose of study treatment.
* Subject has Fridericia-corrected QT interval (QTcF) > 450 msec for males and > 470 msec for females on 12-lead electrocardiogram (ECG) at screening based on local testing.
* Subject has any condition which makes the subject unsuitable for study participation.
* Subject has another active malignancy which is likely to require treatment.
* Subjects who find it difficult to adhere to the provisions of treatment and observation specified in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-10-18 (Actual); Primary Completion 2021-01-22 (Actual); Study Completion 2021-01-22 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) of zolbetuximab: Area under the concentration-time curve (AUC) from the time of dosing extrapolated to time infinity (AUCinf) | Up to 15 months
  AUCinf will be recorded from the PK serum samples collected.
PK of zolbetuximab: Percentage of AUCinf (AUCinf (%extrap)) | Up to 15 months
  AUCinf (%extrap) will be recorded from the PK serum samples collected.
PK of zolbetuximab: AUC from the time of dosing to the last measurable concentration (AUClast) | Up to 15 months
  AUClast will be recorded from the PK serum samples collected.
PK of zolbetuximab: AUC from the time of dosing to the start of the next dosing interval (AUCtau) | Up to 15 months
  AUCtau will be recorded d from the PK serum samples collected.
PK of zolbetuximab: Maximum concertation (Cmax) | Up to 15 months
  Cmax will be recorded from the PK serum samples collected.
PK of zolbetuximab: Concentration immediately prior to dosing at multiple dosing (Ctrough) | Up to 15 months
  Ctrough will be recorded from the PK serum samples collected.
PK of zolbetuximab: Time of the maximum concentration (tmax) | Up to 15 months
  tmax will be recorded from the PK serum samples collected.
PK of zolbetuximab: Terminal elimination half-life (t1/2) | Up to 15 months
  t1/2 will be recorded from the PK serum samples collected.
PK of zolbetuximab: Time of the last measurable concentration (tlast) | Up to 15 months
  tlast will be recorded from the PK serum samples collected.
PK of zolbetuximab: Clearance (CL) | Up to 15 months
  CL will be recorded from the PK serum samples collected.
PK of zolbetuximab: Apparent volume of distribution during the terminal phase (Vz) | Up to 15 months
  Vz will be recorded from the PK serum samples collected.
PK of zolbetuximab: Accumulation ratio calculated using AUC (Rac(AUC)) | Up to 15 months
  Rac(AUC) will be recorded from the PK serum samples collected.
PK of zolbetuximab: Rac (Cmax) | Up to 15 months
  Rac(Cmax)will be recorded from the PK serum samples collected.
Number of participants with adverse events (AEs) | Up to 15 months
  An AE is any untoward medical occurrence in a subject administered a study drug, and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product whether or not considered related to the medicinal product. AE is considered "serious" if the investigator or sponsor view any of the following outcomes: Death, life-threatening, persistent or significant disability/incapacity, congenital anomaly or birth defect, hospitalization, or medically important event. Treatment Emergent Adverse Event (TEAE) is defined as an adverse event observed after starting administration of the study drug and within 30 days after the last dose of study drug.
Number of participants with laboratory test abnormalities and/or AEs | Up to 13 months
  Number of participants with potentially clinically significant laboratory values.
Number of participants with body weight abnormalities and/or AEs | Up to 13 months
  Number of participants with potentially clinically significant body weight changes.
Number of participants with vital sign abnormalities and/or AEs | Up to 13 months
  Number of participants with potentially clinically significant vital sign values.
Number of participants with 12-lead electrocardiogram (ECG) abnormalities and/or AEs | Up to 13 months
  Number of participants with potentially clinically significant 12-ECG values.
Eastern Cooperative Oncology Group (ECOG) performance status score | Up to 13 months
  ECOG performance status will be assessed on the following 6-point scale; 0=Fully active, able to carry on all pre-disease performance without restriction; 1=Restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature, (e.g., light housework, office work); 2=Ambulatory and capable of all self-care, but unable to carry out any work activities. Up and about more than 50% of waking hours; 3=Capable of only limited self-care, confined to bed or chair more than 50% of waking hours; 4=Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair; 5=Dead. Decrease in the score indicates an improvement. Increase in the score indicates a decline in performance.

SECONDARY OUTCOMES:
Proportion of anti-drug antibody (ADA) positive participants | Up to 15 months
  Proportion of participants with presence of ADA will be assessed.
Objective Response Rate (ORR) | Up to 12 months
  ORR is defined as the proportion of subjects whose best overall response (BOR) is rated as compete response (CR) or partial response (PR) among all analyzed subjects. Complete response (CR) of target lesions is defined as disappearance of all target lesions. Any pathological lymph nodes, if chosen as target lesions, must have a reduction in the short axis to < 10 mm from the baseline measurement. Partial response (PR) of target lesions is defined as at least a 30% decrease in the sum of diameters of target lesions (long diameter for non-pathological lymph nodes and short diameter for pathological lymph nodes), taking the baseline sum diameter as a reference. BOR rated as CR or PR should be confirmed by at least 2 consecutive assessments performed at a minimum interval of 4 weeks. Subjects must therefore meet the criteria for CR or PR continuously for 4 weeks or longer.
Duration of Progression Free Survival (PFS) | Up to 12 months
  PFS is defined as the time from the start of study treatment until death from any cause, or radiographic or clinical disease progression per RECIST 1.1, whichever occurs earlier.
Disease Control Rate (DCR) | Up to 12 months
  DCR is defined as the proportion of subjects whose BOR is rated as CR, PR, or stable disease (SD) among all analyzed subjects. SD of target lesions is defined as neither sufficient shrinkage to qualify for PR, nor sufficient increase to qualify for progressive disease (PD), taking the smallest sum diameter on study as a reference. (PD) of the target lesions is defined as at least a 20% increase in the sum of the diameters of target lesions (long diameter for non-pathological lymph nodes and short diameter for pathological lymph nodes), taking the smallest sum on study (this includes the baseline sum if that is the smallest on study) as a reference. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Duration of Response (DOR) | Up to 12 months
  DOR is defined as the time from the date of the first response (CR or PR) per RECIST 1.1 to the date of radiological PD, clinical progression only if radiological assessment is not available, or death, whichever occurs earlier.
Duration of Overall Survival (OS) | Up to 15 months
  OS is defined as the time from the date of randomization until the date of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Science Manager, Study Director — Astellas Pharma China, Inc.
Locations (1):
- Site CN86001, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results and other applicable study documents on the Astellas Clinical Trials website — https://www.clinicaltrials.astellas.com/study/8951-CL-0105/
- See also: Link to plain language summary of the study on the Trial Results Summaries website — https://www.trialsummaries.com/Study/StudyDetails?id=14688&tenant=MT_AST_9011